CLINICAL TRIAL: NCT02664558
Title: A Phase 2, Randomized, Double-BLInd, Placebo- Controlled Study of UBEnimex in Patients With Pulmonary ARTerial HYpertension (WHO Group 1) (LIBERTY)
Brief Title: A Study of Ubenimex in Patients With Pulmonary Arterial Hypertension (WHO Group 1)
Acronym: LIBERTY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIG-UBX-001
Record Dates: First submitted 2016-01-21; First posted 2016-01-27 (Estimated); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ubenimex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ubenimex (Experimental): ubenimex capsules 150 mg three times a day (TID), administered orally for a total of 24 weeks.
  Interventions: Drug: ubenimex
- placebo (Placebo Comparator): placebo capsules TID, administered orally for a total of 24 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ubenimex
  Other Names: UBX
  Arms: ubenimex
Other: placebo
  Arms: placebo

SUMMARY:
This proof-of-concept study is designed as a Phase 2, multicenter, randomized, double-blind, placebo controlled study comparing ubenimex with placebo in patients with pulmonary arterial hypertension (PAH) (World Health Organization [WHO] Group 1) and have a WHO/New York Heart Association (NYHA) Functional Classification (WHO/NYHA-FC) of II or III.

DETAILED DESCRIPTION:
Ubenimex is being developed for the treatment of PAH (WHO Group 1) to improve exercise capacity and delay clinical worsening. This proof-of-concept study is designed as a Phase 2, multicenter, randomized, double-blind, placebo controlled study comparing ubenimex with placebo in patients with PAH (WHO Group 1) and have a WHO/NYHA Functional Classification (WHO/NYHA-FC) of II or III. The Primary Objectives for the study are:

* To evaluate the efficacy of ubenimex in patients with PAH (WHO Group 1).
* To evaluate the safety and tolerability of ubenimex in patients with WHO Group 1 PAH.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 years old.
2. Has a diagnosis of WHO Group 1 PAH.
3. Right heart catheterization performed at Screening with results that are:

   1. Mean pulmonary arterial pressure ≥25 mmHg (at rest) and
   2. Pulmonary venous hypertension (measured as pulmonary capillary wedge pressure (PCWP) ≤15 mmHg. If PCWP is not available, then mean left atrial pressure or left ventricular end-diastolic pressure ≤15 mmHg in the absence of left atrial obstruction. and
   3. Pulmonary vascular resistance (PVR) ≥300 dyn•s/cm5 (3.75 Wood units)
4. Has WHO/NYHA-FC of II or III.
5. Be on stable dose of at least one of the following PAH-specific therapies: endothelin receptor antagonist, an agent acting on the nitric oxide pathway (phosphodiesterase type 5 inhibitor or soluble guanylate cyclase stimulator), and/or a prostacyclin or prostacyclin analog.
6. Has a 6-minute walk distance that is ≥150 and ≤500 meters.
7. Have a ventilation-perfusion scan that rules out thromboembolic disease.

Exclusion Criteria:

Exclusions Related to Cardiovascular Disease

1. History of uncontrolled hypertension
2. Persistent hypotension at Screening.
3. Evidence or history of left-sided heart disease and/or clinically significant cardiac disease in which pulmonary hypertension is more likely WHO Group 2.
4. Acute decompensated heart failure within 1 month of Screening.
5. Recent initiation (<8 weeks from Screening) or planned initiation of cardiopulmonary rehabilitation exercise program.

   Exclusions Related to Pulmonary Disease
6. Newly diagnosed with PAH and not on PAH-specific therapy.
7. Pulmonary hypertension due to:

   1. Uncorrected congenital systemic-to-pulmonary shunt.
   2. Pulmonary veno-occlusive disease and/or pulmonary capillary hemangiomatosis
   3. Persistent pulmonary hypertension of the newborn
   4. WHO clinical classification Groups 2-5
8. Evidence of significant airway and/or parenchymal lung disease.
9. Chronic infection related to tuberculosis or fungal or mycobacterial disease.

   Exclusions Based on Other Medical Conditions
10. Chronic infections including, but not limited to tuberculosis (TB), hepatitis B virus (HBV) or hepatitis C virus (HCV).
11. History of portal hypertension or chronic liver disease, including positive serology for infection with HCV and/or HBV.
12. Evidence of active infection requiring intravenous or oral antibiotics within 4 weeks of Screening.
13. Body mass index ≥35.0 at Screening.
14. History of obstructive sleep apnea.
15. History of malignancy within the last 5 years, except nonmelanoma skin cancer and cervical carcinoma in situ treated with curative intent.
16. Neuropsychiatric disorders/symptoms or psychological conditions.
17. Pregnancy or breast-feeding
18. Prior treatment with B cell or lymphocyte-depleting agents (eg, rituximab, Campath)

    Exclusions Based on Concomitant Medication Use
19. Concurrent regular use of another leukotriene pathway inhibitor, including over-the-counter medications or herbal remedies.

    Exclusions Based on Laboratory Values
20. Significant/chronic renal insufficiency.
21. Transaminases (alanine transaminase, aspartate transaminase) levels >3 × upper limit of normal (ULN) and/or bilirubin level >2 × ULN.
22. Absolute neutrophil count <1500 mm3.
23. Hemoglobin concentration <9 g/dL at Screening.
24. Hepatic dysfunction as defined by Child-Pugh Class B or C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-04; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Heart Center Foundation, An Affiliate of Cedars-Sinai Heart Institute, Cedars-Sinai Medical Care Foundation, Beverly Hills, California
  - UCSD Medical Center, La Jolla, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Cleveland Clinic, Florida, Weston, Florida
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Chest Medicine Associates, South Portland, Maine
  - Johns Hopkins University, Pulmonary and Critical Care Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Weill Cornell Medicine, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Respiratory Institute, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pennsylvania Medical Center, Pittsburgh, Pennsylvania
  - Alpert Medical School of Brown University Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University Texas Health Science Center, San Antonio, Texas
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Tian W, Jiang X, Tamosiuniene R, Sung YK, Qian J, Dhillon G, Gera L, Farkas L, Rabinovitch M, Zamanian RT, Inayathullah M, Fridlib M, Rajadas J, Peters-Golden M, Voelkel NF, Nicolls MR. Blocking macrophage leukotriene b4 prevents endothelial injury and reverses pulmonary hypertension. Sci Transl Med. 2013 Aug 28;5(200):200ra117. doi: 10.1126/scitranslmed.3006674. PMID 23986401
- [Background] Qian J, Tian W, Jiang X, Tamosiuniene R, Sung YK, Shuffle EM, Tu AB, Valenzuela A, Jiang S, Zamanian RT, Fiorentino DF, Voelkel NF, Peters-Golden M, Stenmark KR, Chung L, Rabinovitch M, Nicolls MR. Leukotriene B4 Activates Pulmonary Artery Adventitial Fibroblasts in Pulmonary Hypertension. Hypertension. 2015 Dec;66(6):1227-1239. doi: 10.1161/HYPERTENSIONAHA.115.06370. Epub 2015 Oct 5. PMID 26558820

RESULTS

PARTICIPANT FLOW:
Groups:
- Ubenimex: ubenimex capsules 150 mg three times a day (TID), administered orally for a total of 24 weeks.
  ubenimex
- Placebo: placebo capsules TID, administered orally for a total of 24 weeks
  placebo
Period: Overall Study
Arm/Group | Ubenimex | Placebo
Started | 41 | 20
Completed | 36 | 18
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ubenimex | Placebo | Total
Number analyzed (Participants) | 41 | 20 | 61
Age, Continuous [Mean (Full Range); unit: years] | 49.9 [18 to 75] | 53.0 [18 to 75] | 50.9 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 15 | 51
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 18 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Mean pulmonary vascular resistance (PVR) [Mean (Standard Deviation); unit: dyn•s/cm^5] — PVR was assessed by hemodynamic measurements obtained via right heart catheterization.
  dyn•s/cm^5 | 649.9 (315.8) | 624.4 (217.1) | 641.57 (217.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Vascular Resistance (PVR)
Description: Change from Baseline at End of Treatment in PVR Using Worst Case Imputation in the Modified Intent to Treat Population. PVR was assessed by hemodynamic measurements obtained via right heart catheterization.
Time Frame: Baseline to Week 24
Population: Modified Intent to Treat Population: i.e., all randomized patients who received at least one dose of study drug and had a baseline assessment for the respective endpoint.
Measure: Mean (Standard Deviation); unit: dyn.sec/cm5
Arm/Group | Ubenimex | Placebo
Number analyzed (Participants) | 41 | 20
dyn.sec/cm5 | 73.1 (271.6) | 46.6 (256.8)

2. Secondary Outcome: Change in 6-minute Walk Distance (6MWD)
Description: Change in exercise capacity from baseline to Week 24 as determined by the 6MWD
Time Frame: Baseline to Week 24
Population: Modified intention-to-treat population: i.e., all randomized patients who received at least one dose of study drug and had a baseline assessment for the respective endpoint.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Ubenimex | Placebo
Number analyzed (Participants) | 41 | 20
meters | -20.0 (12.79) | 4.2 (17.38)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Ubenimex | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/20
Serious Adverse Events (participants affected / at risk) | 9/41 | 2/20
Other Adverse Events (participants affected / at risk) | 39/41 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ubenimex (N=41) | Placebo (N=20)
Complication associated with device (General disorders) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Diarrhoea infectious (General disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Progressive pulmonary hypertension (Reproductive system and breast disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ubenimex (N=41) | Placebo (N=20)
Diarrhea (Gastrointestinal disorders) | 11 | 5
Nausea (Gastrointestinal disorders) | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Headache (Nervous system disorders) | 5 | 6
Hypokalemia (Metabolism and nutrition disorders) | 5 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT02664558/Prot_SAP_000.pdf